CLINICAL TRIAL: NCT06546267
Title: Efficacy of Advanced Radiotherapy (ART) in Prostate Cancer Patients With Early Stage, Advanced, Metastatic and Relapsed Disease (PROST-ART)
Brief Title: Advanced Radiotherapy (ART) in Prostate Cancer (PROST-ART)
Acronym: PROST-ART
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Nadia Di Muzio, Professor, IRCCS San Raffaele
Other Study IDs: PROST-ART
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Radiotherapy; Adjuvant Radiotherapy; Salvage Radiotherapy; Stereotactic Body Radiotherapy (SBRT); Simultaneous Integrated Boost; Oligometastatic Disease; Bone Metastases; Lymph-Node Metastases; Choline PET/CT; PSMA PET/CT; PET guidance
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prostate cancer, localized disease: Patients treated with IGRT, IMRT, SBRT, with radical intent for localized prostate cancer will be evaluated
  Other Names:
  Intensity Modulated Radiotherapy Stereotactic Body Radiotherapy
  Interventions: Radiation: Image Guided Radiotherapy; Radiation: Intensity Modulated Radiotherapy; Radiation: Stereotactic Body Radiotherapy
- Prostate cancer, extensive disease: Patients operated on for prostate cancer, treated with IGRT, IMRT, SBRT in adjuvant setting will be evaluated
  Other Names:
  Intensity Modulated Radiotherapy Stereotactic Body Radiotherapy
  Interventions: Radiation: Image Guided Radiotherapy; Radiation: Intensity Modulated Radiotherapy; Radiation: Stereotactic Body Radiotherapy
- Prostate cancer, biochemical relapse: Patients operated on for prostate cancer and treated with IGRT, IMRT, SBRT for biochemical relapse will be evaluated
  Interventions: Radiation: Image Guided Radiotherapy; Radiation: Intensity Modulated Radiotherapy; Radiation: Stereotactic Body Radiotherapy
- Prostate cancer, oligometastatic disease ( lymph-nodal, bone, visceral): Prostate cancer patients treated with IGRT, IMRT, SBRT, in radical setting or as salvage radiotherapy for relapse after previous treatments will be evaluated
  Interventions: Radiation: Image Guided Radiotherapy; Radiation: Intensity Modulated Radiotherapy; Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Image Guided Radiotherapy — Patients treated with IGRT for Prostate cancer will be evaluated
  Other Names: IGRT
Radiation: Intensity Modulated Radiotherapy — Patients treated with IMRT for Prostate cancer will be evaluated
  Other Names: IMRT
Radiation: Stereotactic Body Radiotherapy — Patients treated with SBRT for Prostate cancer will be evaluated
  Other Names: SBRT, SRT, SABR (Stereotactic Ablative Radiotherapy)

SUMMARY:
This is a retrospective monoinstitutional study which analyses the results of advanced radiotherapy (IGRT, IMRT, SBRT, and PET-guided) performed for radical, adjuvant, or salvage purposes in patients with low, intermediate, high, and very high-risk prostate cancer, or with biochemical, lymph node, or oligometastatic recurrence treated between 2004 and 2024.

Approved by Ethics Committee of IRCCS San Raffaele Hospital Approval Number: 187/INT/2021, 03/02/2022

Amendment approved by Ethics Committee 1, Lombardy Region Approval number CET Em. 194-2024, 22/05/2024

DETAILED DESCRIPTION:
This is a single-center, retrospective study (PROST-ART) that has as its primary objective the evaluation of the efficacy of radiotherapy treatments performed in patients with early-stage, advanced, metastatic prostate disease, with biochemical relapses after surgery, with local relapses after radiotherapy, or oligometastatic/oligoprogressive disease. The aim of the study is to measure the biochemical relapse-free survival (bRFS), local and regional relapse (LR, regional relapse, RR), distant metastases-free survival (DMS), clinical relapse (DFS), disease-free survival (PCSS), and overall survival (OS) from both disease diagnosis and the end of radiotherapy until the last useful follow-up, or until the patient's death. In addition, the acute and late toxicity of treatments will be assessed from the start of treatment until the last follow-up/death of the patient and the period without other oncological treatments, from the end of treatment until the start of another oncological treatment/last follow-up.

At least 200 patients treated in the last 5 years, some receiving stereotactic radiotherapy to the prostate, or prostate and seminal vesicles, and the others pelvic lymph node and prostate irradiation, who are still alive and contactable, and agree to participate, will be included in a survey on quality of life (QoL). These patients, after signing an informed consent for the collection of new information, will receive an EORTC QLQ-PR25 quality of life questionnaire, in order to quantify the impact of toxicity. In addition, the radiomic characteristics of the computed tomography/ PET-CT performed for treatment planning along with evaluation of the results will be extracted to identify related predictive factors.

The QoL study is configured as retrospective as the questionnaire will only be an expression, from the patient's point of view, of the toxicity of the previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients, > 18 years old, treated with IGRT, IMRT, SBRT

Exclusion Criteria:

* other tumors
* > 95 years old

Ages: 18 Years to 95 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer
Study Population: Prostate cancer patients with early-stage, advanced, metastatic prostate disease, with biochemical relapses after surgery, with local relapses after radiotherapy, or oligometastatic/oligoprogressive disease (lymph nodes, bone, visceral)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Local Relapse Free Survival | From the date of radiotherapy end until the date of local progression or date of death from any cause, whichever came first, assessed up to 120 months
  Local control of the disease (at the treated site)
Regional Relapse Free Survival | From the date of radiotherapy end until the date of regional progression or date of death from any cause, whichever came first, assessed up to 120 months
  Regional control of the disease (at the regional lymph node chain)
Distant Metastasis Free Survival | From the date of radiotherapy end until the date of distant progression or date of death from any cause, whichever came first, assessed up to 120 months
  Distant Metastasis developed after the treatment
Biochemical relapse free survival | From the date of radiotherapy end until the date of biochemical progression or date of death from any cause, whichever came first, assessed up to 120 months
  Biochemical relapse after the treatment
Disease Free Survival | From the date of radiotherapy end until the date of first documented clinical progression or date of death from any cause, whichever came first, assessed up to 120 months
  Absence of disease progression during the follow-up
Overall Survival | From the date of radiotherapy end until the date of death from any cause, assessed up to 120 months
  Survival from all causes
Cancer Specific Survival | From the date of radiotherapy end until the date of death from disease progression, assessed up to 120 months
  Cancer Survival

SECONDARY OUTCOMES:
Acute Toxicity | Up to three months from the start of radiotherapy
  Toxicity developed in the first three months after the treatment, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity
Late toxicity | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 120 months
  Toxicity developed after three months until the end of follow-up or death, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity

OTHER OUTCOMES:
Predictive factors for disease progression and death | From radiotherapy end to date of local, regional progression, distant failure, or death, assessed up to 120 months
  Factors predicting survival. Survival trees, univariate/multivariate Cox regression models will be estimated to identify potential risk factors associated with survival outcomes
Radiomic predictive factors for disease progression and death | From radiotherapy end to the first registered event (disease progression or death), assessed up to 120 months
  CT and PET/CT radiomic features predicting relapse or death will be extracted, acording to IBSI (Image Biomarker Standardisation Initiative), owning to the different families of features: Morphology, Statistical, Intensity Histogram, Grey Level Cooccurrence Matrix 3D-average, Grey Level Co-occurrence Matrix 3D-combined, Grey Level Run Lenght 3D-average. Grey Level Run Lenght 3D_combined, Grey Level Size Zone Matrix 3D, Neighbors Grey Tone Difference Matrix 3D, Grey Level Distance Zone Matrix 3D, standard convolutional filters within radiomic workflow (wavelets, Laplacian of Gaussian)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Di Muzio, Prof, Principal Investigator — IRCCS San Raffaele, Milan
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author (AF) will be evaluated by the Lombardy Territorial Ethics Committee 1.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for another 2 years after the closure of the study
Access Criteria: Request from the corresponding author approved by the Lombardy Territorial Ethics Committee 1

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Result] Parker CC, James ND, Brawley CD, Clarke NW, Hoyle AP, Ali A, Ritchie AWS, Attard G, Chowdhury S, Cross W, Dearnaley DP, Gillessen S, Gilson C, Jones RJ, Langley RE, Malik ZI, Mason MD, Matheson D, Millman R, Russell JM, Thalmann GN, Amos CL, Alonzi R, Bahl A, Birtle A, Din O, Douis H, Eswar C, Gale J, Gannon MR, Jonnada S, Khaksar S, Lester JF, O'Sullivan JM, Parikh OA, Pedley ID, Pudney DM, Sheehan DJ, Srihari NN, Tran ATH, Parmar MKB, Sydes MR; Systemic Therapy for Advanced or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Radiotherapy to the primary tumour for newly diagnosed, metastatic prostate cancer (STAMPEDE): a randomised controlled phase 3 trial. Lancet. 2018 Dec 1;392(10162):2353-2366. doi: 10.1016/S0140-6736(18)32486-3. Epub 2018 Oct 21. PMID 30355464
- [Result] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Result] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Result] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Result] Incrocci L, Wortel RC, Alemayehu WG, Aluwini S, Schimmel E, Krol S, van der Toorn PP, Jager H, Heemsbergen W, Heijmen B, Pos F. Hypofractionated versus conventionally fractionated radiotherapy for patients with localised prostate cancer (HYPRO): final efficacy results from a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1061-1069. doi: 10.1016/S1470-2045(16)30070-5. Epub 2016 Jun 20. PMID 27339116
- [Result] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Result] Pollack A, Walker G, Horwitz EM, Price R, Feigenberg S, Konski AA, Stoyanova R, Movsas B, Greenberg RE, Uzzo RG, Ma C, Buyyounouski MK. Randomized trial of hypofractionated external-beam radiotherapy for prostate cancer. J Clin Oncol. 2013 Nov 1;31(31):3860-8. doi: 10.1200/JCO.2013.51.1972. Epub 2013 Oct 7. PMID 24101042
- [Result] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373
- [Result] Parker CC, Clarke NW, Cook AD, Kynaston HG, Petersen PM, Catton C, Cross W, Logue J, Parulekar W, Payne H, Persad R, Pickering H, Saad F, Anderson J, Bahl A, Bottomley D, Brasso K, Chahal R, Cooke PW, Eddy B, Gibbs S, Goh C, Gujral S, Heath C, Henderson A, Jaganathan R, Jakobsen H, James ND, Kanaga Sundaram S, Lees K, Lester J, Lindberg H, Money-Kyrle J, Morris S, O'Sullivan J, Ostler P, Owen L, Patel P, Pope A, Popert R, Raman R, Roder MA, Sayers I, Simms M, Wilson J, Zarkar A, Parmar MKB, Sydes MR. Timing of radiotherapy after radical prostatectomy (RADICALS-RT): a randomised, controlled phase 3 trial. Lancet. 2020 Oct 31;396(10260):1413-1421. doi: 10.1016/S0140-6736(20)31553-1. Epub 2020 Sep 28. PMID 33002429
- [Result] Kneebone A, Fraser-Browne C, Duchesne GM, Fisher R, Frydenberg M, Herschtal A, Williams SG, Brown C, Delprado W, Haworth A, Joseph DJ, Martin JM, Matthews JHL, Millar JL, Sidhom M, Spry N, Tang CI, Turner S, Wiltshire KL, Woo HH, Davis ID, Lim TS, Pearse M. Adjuvant radiotherapy versus early salvage radiotherapy following radical prostatectomy (TROG 08.03/ANZUP RAVES): a randomised, controlled, phase 3, non-inferiority trial. Lancet Oncol. 2020 Oct;21(10):1331-1340. doi: 10.1016/S1470-2045(20)30456-3. PMID 33002437
- [Result] Vale CL, Fisher D, Kneebone A, Parker C, Pearse M, Richaud P, Sargos P, Sydes MR, Brawley C, Brihoum M, Brown C, Chabaud S, Cook A, Forcat S, Fraser-Browne C, Latorzeff I, Parmar MKB, Tierney JF; ARTISTIC Meta-analysis Group. Adjuvant or early salvage radiotherapy for the treatment of localised and locally advanced prostate cancer: a prospectively planned systematic review and meta-analysis of aggregate data. Lancet. 2020 Oct 31;396(10260):1422-1431. doi: 10.1016/S0140-6736(20)31952-8. Epub 2020 Sep 28. PMID 33002431
- [Result] Ost P, Reynders D, Decaestecker K, Fonteyne V, Lumen N, De Bruycker A, Lambert B, Delrue L, Bultijnck R, Claeys T, Goetghebeur E, Villeirs G, De Man K, Ameye F, Billiet I, Joniau S, Vanhaverbeke F, De Meerleer G. Surveillance or Metastasis-Directed Therapy for Oligometastatic Prostate Cancer Recurrence: A Prospective, Randomized, Multicenter Phase II Trial. J Clin Oncol. 2018 Feb 10;36(5):446-453. doi: 10.1200/JCO.2017.75.4853. Epub 2017 Dec 14. PMID 29240541
- [Result] Di Muzio NG, Fodor A, Noris Chiorda B, Broggi S, Mangili P, Valdagni R, Dell'Oca I, Pasetti M, Deantoni CL, Chiara A, Berardi G, Briganti A, Calandrino R, Cozzarini C, Fiorino C. Moderate Hypofractionation with Simultaneous Integrated Boost in Prostate Cancer: Long-term Results of a Phase I-II Study. Clin Oncol (R Coll Radiol). 2016 Aug;28(8):490-500. doi: 10.1016/j.clon.2016.02.005. Epub 2016 Mar 5. PMID 26961088
- [Result] Cozzarini C, Fiorino C, Di Muzio N, Alongi F, Broggi S, Cattaneo M, Montorsi F, Rigatti P, Calandrino R, Fazio F. Significant reduction of acute toxicity following pelvic irradiation with helical tomotherapy in patients with localized prostate cancer. Radiother Oncol. 2007 Aug;84(2):164-70. doi: 10.1016/j.radonc.2007.07.013. Epub 2007 Aug 13. PMID 17706308
- [Result] Fodor A, Fiorino C, Picchio M, Di Muzio N. Re: Daniel E. Spratt, Herbert A. Vargas, Zachary S. Zumsteg, et al. Patterns of Lymph Node Failure after Dose-escalated Radiotherapy: Implications for Extended Pelvic Lymph Node Coverage. Eur Urol 2017;71;37-43: High-dose Radiotherapy and Pelvic Lymph Nodal Irradiation for High-risk Prostate Cancer in the Image-guided Radiotherapy Era. Eur Urol. 2017 Jun;71(6):e179-e180. doi: 10.1016/j.eururo.2016.12.021. Epub 2017 Jan 5. No abstract available. PMID 28065538
- [Result] Di Muzio N, Fiorino C, Cozzarini C, Alongi F, Broggi S, Mangili P, Guazzoni G, Valdagni R, Calandrino R, Fazio F. Phase I-II study of hypofractionated simultaneous integrated boost with tomotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Jun 1;74(2):392-8. doi: 10.1016/j.ijrobp.2008.08.038. Epub 2008 Dec 4. PMID 19056184
- [Result] Fiorino C, Di Muzio N, Broggi S, Cozzarini C, Maggiulli E, Alongi F, Valdagni R, Fazio F, Calandrino R. Evidence of limited motion of the prostate by carefully emptying the rectum as assessed by daily MVCT image guidance with helical tomotherapy. Int J Radiat Oncol Biol Phys. 2008 Jun 1;71(2):611-7. doi: 10.1016/j.ijrobp.2008.01.048. Epub 2008 Apr 18. PMID 18374511
- [Result] Cozzarini C, Fiorino C, Deantoni C, Briganti A, Fodor A, La Macchia M, Noris Chiorda B, Rancoita PM, Suardi N, Zerbetto F, Calandrino R, Montorsi F, Di Muzio N. Higher-than-expected severe (Grade 3-4) late urinary toxicity after postprostatectomy hypofractionated radiotherapy: a single-institution analysis of 1176 patients. Eur Urol. 2014 Dec;66(6):1024-30. doi: 10.1016/j.eururo.2014.06.012. Epub 2014 Jun 27. PMID 24985964
- [Result] Fodor A, Berardi G, Fiorino C, Picchio M, Busnardo E, Kirienko M, Incerti E, Dell'Oca I, Cozzarini C, Mangili P, Pasetti M, Calandrino R, Gianolli L, Di Muzio NG. Toxicity and efficacy of salvage carbon 11-choline positron emission tomography/computed tomography-guided radiation therapy in patients with lymph node recurrence of prostate cancer. BJU Int. 2017 Mar;119(3):406-413. doi: 10.1111/bju.13510. Epub 2016 May 24. PMID 27104782
- [Result] Deantoni CL, Fodor A, Cozzarini C, Fiorino C, Brombin C, Di Serio C, Calandrino R, Di Muzio N. Prostate cancer with low burden skeletal disease at diagnosis: outcome of concomitant radiotherapy on primary tumor and metastases. Br J Radiol. 2020 Apr;93(1108):20190353. doi: 10.1259/bjr.20190353. Epub 2020 Jan 31. PMID 31971828